CLINICAL TRIAL: NCT00472017
Title: Phase I Trial of Vandetanib (ZD6474, ZACTIMA) With Concurrent Radiation in Treatment of Newly Diagnosed Brainstem Glioma
Brief Title: Vandetanib and Radiation Therapy in Treating Young Patients With Newly Diagnosed Diffuse Brainstem Glioma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SJBG07-SJ
Record Dates: First submitted 2007-05-08; First posted 2007-05-10 (Estimated); Last update posted 2012-10-15 (Estimated); Status verified 2012-10

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: untreated childhood brain stem glioma
MeSH Terms: conditions — Central Nervous System Neoplasms | interventions — vandetanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pediatric Diffuse Brainstem Glioma Patients (Experimental): Patients with newly diagnosed diffuse brainstem gliomas receive vandetanib.
  Interventions: Drug: vandetanib

INTERVENTIONS:
Drug: vandetanib — Oral vandetanib administration will start on the same day as RT. Treatment with vandetanib will extend for the entire duration of RT, and then will be continued after completion of RT for a maximum duration of 2 years.
  Other Names: ZD6474; Zactima

SUMMARY:
This phase I trial is studying the side effects and best dose of vandetanib when given together with radiation therapy in treating young patients with newly diagnosed diffuse brain stem glioma.

DETAILED DESCRIPTION:
Vandetanib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Specialized radiation therapy that delivers a high dose of radiation directly to the tumor may kill more tumor cells and cause less damage to normal tissue. Giving vandetanib together with radiation therapy may kill more tumor cells.

Patients undergo conformal radiotherapy once daily, 5 days a week, for 6 weeks. Patients also receive oral vandetanib once daily beginning on the same day as radiotherapy and continuing for up to 2 years in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of vandetanib until the maximum tolerated dose (MTD) is determined.

Blood samples are collected periodically for pharmacokinetic studies, polymorphism analysis (e.g., CYP3A4/5), and immunological laboratory methods (e.g., western blot assay). Imaging studies are also conducted periodically.

ELIGIBILITY:
* Diagnosis of 1 of the following:

  * Diffuse brainstem glioma
  * High-grade glioma originating from brainstem
* Age must be greater than or equal to 2 years and less than 21 years
* Newly diagnosed disease
* Lansky OR Karnofsky performance status 40-100%
* ANC ≥ 1,000/mm³
* Platelet count ≥ 100,000/mm³ (transfusion independent)
* Hemoglobin ≥ 8 g/dL (transfusion allowed)
* Bilirubin < 1.5 times upper limit of normal (ULN) for age
* ALT < 5 times ULN
* Albumin ≥ 2 g/dL
* Creatinine < 2 times ULN for age OR glomerular filtration rate > 70 mL/min
* QTc interval < 450 msec by EKG
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

Ages: 2 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 35 (Actual)
Dates: Start 2007-04; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
To estimate the maximum tolerated dose (MTD) and to determine the dose-limiting toxicity (DLT) of vandetanib administered concurrently with radiation therapy (RT) in pediatric patients with newly diagnosed diffuse brainstem glioma. | 3 Years

SECONDARY OUTCOMES:
To determine the toxicities associated with the chronic use of vandetanib in pediatric patients | 3 Years
To characterize the pharmacokinetics of vandetanib in pediatric patients | 3 Years
To evaluate the influence of specific polymorphisms on the pharmacokinetics of vandetanib in children | 3 Years
To prospectively investigate the role of innovative imaging techniques (e.g., perfusion/diffusion, susceptibility-weighted imaging, arterial spin labeling) in assessing the response to therapy, particularly in tumor vascularization and perfusion | 3 Years
To prospectively estimate the cumulative incidence of intratumoral hemorrhage in patients with diffuse brainstem glioma treated with vandetanib concurrently with and after RT in the context of a Phase I study | 3 Years
Prospectively assess the number of circulating endothelial cells and circulating endothelial progenitors before the start and during therapy and, if possible, to correlate these findings with tumor response, imaging studies, and other biological assays | 3 Years

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Broniscer, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org